CLINICAL TRIAL: NCT05503966
Title: Combining Antidepressants and Attention Bias Modification in Depression: a Randomized Controlled Trial in Primary Care
Brief Title: Combining Antidepressants and Attention Bias Modification in Depression
Acronym: DEPTREAT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oslo (Other)
Collaborators: University of Oxford (Other)
Responsible Party: Principal Investigator, Jan Ivar Rossberg, Professor, University of Oslo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 273292
Record Dates: First submitted 2022-08-09; First posted 2022-08-17 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2024-05

CONDITIONS: Depressive Disorder
Keywords: Major Depressive Disorder; Attentional Bias Modification; Primary Health Care
MeSH Terms: conditions — Depressive Disorder; Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: The study is a three-armed, double-blinded, pragmatic randomized controlled trial comparing the efficacy of ABM as add-on to treatment with antidepressants (SSRI ABM group) in primary care compared to standard antidepressant treatment (SSRI TAU group). The third group will in addition to TAU be engaged in answering all the questionnaires and perform all the tasks, but without ABM, thus controlling for being engaged in some cognitive activity (SSRI Active comparison group).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Positive ABM (Experimental): The ABM intervention will be initiated two weeks after antidepressant treatment started (baseline) and continues with two daily sessions for two weeks.
  Interventions: Behavioral: Attentional Bias Modification
- No ABM (Active Comparator): This group will in addition to TAU complete the schedule of intermediate assessments as in the ABM group, but no ABM , thus controlling for the aspects of the ABM group that are additional to TAU (increased engagement in cognitive activity and repeated assessment over time), but not including the training component itself (SSRI Active comparison group).
  Interventions: Behavioral: Attentional Bias Modification
- TAU (No Intervention): Patients allocated to this group will be assessed at baseline and at the primary end-point as well after 12 weeks and 6 months follow-up. They will not complete any instruments during the intervention period to prevent the effect of some cognitive activity and provide a more ecologically valid version of TAU as it happens in primary care.

INTERVENTIONS:
Behavioral: Attentional Bias Modification — The ABM task is based on a computerized visual Dot-probe task. In the dot-probe task paired stimuli of negative (angry and fearful), positive (happy) or neutral faces are presented, followed by one or two probes (dots) appearing in the spatial location of one of the stimuli. Participants are then required to press one of two buttons as quickly as possible to indicate the number of dots in the probe. In the ABM condition, probes are in the same locus as the more positive/less negative stimuli in 87% of the trials, as opposed to 13% with probes in the same locus as more negative/less positive stimuli. Thus, when completing the ABM, participants should learn to deploy their attention toward the relatively more positive stimuli, and in this way develop a more positive AB.
  Other Names: ABM
  Arms: No ABM; Positive ABM

SUMMARY:
Background: Major depressive disorder (MDD) is a highly prevalent psychiatric condition associated with significant disability, mortality and economic burden. A large proportion of MDD patients are treated in primary health care (PHC) in the municipalities and represent a challenging group. Attentional Bias Modification (ABM) training in combination with antidepressants (SSRIs) could be an effective treatment. The overall aim of this study is to test the hypothesis that adding an ABM procedure to regular treatment with antidepressants in PHC will result in further improvement of symptoms compared to treatment with antidepressants alone (treatment as usual, TAU) and as compared to an active comparison condition.

Methods: A total of 246 patients with a diagnosis of MDD will be included in this study. The study is a three-armed pragmatic randomized controlled trial comparing the efficacy of ABM as add-on to treatment with antidepressants in primary care (ABM condition) compared to standard antidepressant treatment (TAU condition). In a third group participants will complete the same schedule of intermediate assessments as the ABM condition in addition to TAU , but no ABM, thus controlling for the non-training-specific aspects of the ABM condition (SSRI Active comparison group).

Discussion:

The clinical outcome of this study may help develop easy accessible, low cost treatment of depression in PHC. Moreover, the study aims to broaden our knowledge of optimal treatment for patients with a MDD by providing adjunct treatment to facilitate recovery and long term gain

DETAILED DESCRIPTION:
Major Depressive Disorder (MDD) is a debilitating disorder that affects 15% of the population and is a leading cause of disability worldwide. The economic burden of MDD is enormous, with estimates of direct/indirect costs of $210.2 billion/year in the US alone.

Although both psychotherapy and antidepressant medications are effective, it is not uncommon for a patient with MDD to have temporary symptom reduction after treatment but require an extended amount of time for full restoration of function. A large proportion of MDD patients are treated in PHC in the municipalities and represent a challenging group to treat effectively. At the same time, it is known that early treatment and coordinated follow-up can be efficient even without costly specialist interventions or hospital treatment. Thus, improved treatment of MDD in municipalities represents a tremendous opportunity for improvement of public health and well being in the general population.

Considerable progress has been made in characterizing mechanisms underlying depression vulnerability and this may be harnessed to improve future treatment strategies. The ability to deal effectively with stress and life events is influenced by the ability of the brain to rapidly adapt, which in turn is a function of synaptic plasticity. Further, it has been hypothesized that the capacity of synapses for functional and structural change plays an important role in the pathophysiology and treatment of mood disorders. These dysfunctional neural mechanisms are affected by antidepressants and increased synaptic plasticity may be one of the therapeutic mechanisms. However, enhancing plasticity alone may not lead to a sufficient treatment response in all individuals affected by depression. Indeed, the entrenched attentional biases seen in depression, such as the tendency to focus on and recall negative information, may persist and be further entrenched by changes in the neural underpinnings of learning and memory. Furthermore, negative attention biases are associated with persistence of sad mood in major depressive disorder. However, selective biases in attention can potentially be modified by a simple computerized technique: The Attention Bias Modification Task (ABM).

While some studies have reported an effect of ABM in depression, definitive conclusions have been limited by small samples and poor trial methodology in many studies. However, recently a large RCT study showed that ABM training led to significantly greater decrease in clinician-rated symptoms of depression as compared to the control condition. ABM induced a change in AB towards relatively more positive stimuli for participants that also showed greater symptom reduction. A secondary network analysis indicated that ABM primarily influenced the symptom "interest" which could mediate both symptoms, social support, functioning and quality of life. Furthermore, a sub-sample was included in a brain imaging study revealing that the ABM active group showed reduced activation in the amygdala and the anterior cingulate cortex when passively viewing negative images compared to the sham group. Other studies have also found that experimentally modifying negatively biased attention reduces depressive symptoms. However, some studies have showed that ABM is not significantly better in improving depressive symptoms as compared to sham.

In addition to explore mechanisms of neuroplasticity, in parallel research there has also been interest in understanding the effects of antidepressant drugs on psychological processes involved in depression. Thus, a number of studies for more than a decade have documented that SSRIs modify biases in emotional processing, thus they work by modifying the same underlying basic mechanism that are the focus when applying ABM procedures. Emotional processing is influenced early in the treatment and independently of change in subjective mood, and these effects have been shown in depressed subjects as well as in healthy volunteers. Most of these studies investigated the effects of a single dose of an SSRI compared with placebo. However, it has been showed that antidepressants as prescribed in the community also increases processing for positive information.

A logical next step is to combine SSRIs as prescribed in primary health with an ABM procedure. Combining pharmacological and psychological regimes are gold standard treatment options in both depression and anxiety and is not associated with baseline severity.Treatments, such as cognitive behavioral therapy (CBT) might also change attentional biases, but by implementing an ABM procedure we will more readily target these biases directly. By combining ABM with today's treatment options, we could potentially increase treatment efficacy and shorten treatment duration. Furthermore, ABM has the advantage of being entirely deliverable on a digital platform without the need for therapist interaction.

The main aim of this study is to test the hypothesis that adding an ABM procedure to regular treatment with antidepressants in PHC will result in a clinically important improvement of symptoms compared to treatment with antidepressants alone (TAU), and as compared to an active comparison condition. Secondary aims are to investigate possible effects of the combined treatment on anxiety symptoms, emotional blunting, rumination, perceived stress, psychosocial functioning/work and suicidal risk. Thirdly, a number of potential moderators will also be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Major Depressive Disorder
* BDI II > 14
* Age 18 - 65 years
* Ability to understand and speak a Scandinavian language
* Willingness and ability to give informed consent

Exclusion Criteria:

* Current or past neurological illness
* Traumatic brain injury
* Current alcohol and/or substance dependency disorders
* Psychotic disorders
* Bipolar disorder type 1,
* Developmental disorders and mental retardation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Estimated)
Dates: Start 2022-09-22 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale | 8 weeks after baseline.
  Clinician rated depressive symptoms. Range (0-50). Higher score indicate more depressive symptoms
Beck Depression Inventory II | 8 weeks after baseline.
  Self rated depressive symptoms. Range (0-63). Higher score indicate more depressive symptoms

SECONDARY OUTCOMES:
Beck Depression Inventory II | Follow-up 12 weeks after baseline.
  Self rated depressive symptoms, Range (0-63). Higher score indicate more depressive symptoms
Beck Depression Inventory II | Follow-up 6 months after baseline
  Self rated depressive symptoms, Range (0-63). Higher score indicate more depressive symptoms
Generalized Anxiety Disorder-7 | 8 weeks after baseline.
  Self rated anxiety symptoms. Range (0-21). Higher score indicate more anxiety symptoms
Generalized Anxiety Disorder-7 | 12 weeks after baseline.
  Self rated anxiety symptoms. Range (0-21). Higher score indicate more anxiety symptoms
Generalized Anxiety Disorder-7 | 6 months after baseline
  Self rated anxiety symptoms. Range (0-21). Higher score indicate more anxiety symptoms
Oxford Depression Questionnaire | 8 weeks after baseline
  Self rated emotional blunting symptoms. Range (0-80). Higher score indicate more symptoms.
Oxford Depression Questionnaire | 12 weeks after baseline.
  Self rated emotional blunting symptoms. Range (0-80). Higher score indicate more symptoms.
Oxford Depression Questionnaire | 6 months after baseline
  Self rated emotional blunting symptoms. Range (0-80). Higher score indicate more symptoms.
Rumination Response Scale | 8 weeks after baseline.
  Self rated level of rumination. Range (22-88). Higher score indicate more rumination.
Rumination Response Scale | 12 weeks after baseline
  Self rated level of rumination. Range (22-88). Higher score indicate more rumination.
Rumination Response Scale | 6 months after baseline
  Self rated level of rumination. Range (22-88). Higher score indicate more rumination.
The Perceived Stress Scale | 8 after baseline
  Self rated subjective level of stress. Range (0-40). Higher score indicate more perceived stress.
The Perceived Stress Scale | 12 weeks after baseline
  Self rated subjective level of stress. Range (0-40). Higher score indicate more perceived stress.
The Perceived Stress Scale | 6 months after baseline
  Self rated subjective level of stress. Range (0-40). Higher score indicate more perceived stress.
The Work and Social Adjustment Scale | 8 weeks after baseline.
  Self rated level of social functioning. Range (0-40). Higher score indicate poorer functioning
The Work and Social Adjustment Scale | 12 weeks after baseline.
  Self rated level of social functioning. Range (0-40). Higher score indicate poorer functioning
The Work and Social Adjustment Scale | 6 months after baseline.
  Self rated level of social functioning. Range (0-40). Higher score indicate poorer functioning
Bergen Insomnia Scale | 8 weeks after baseline.
  Self rated level of sleep problems. Range (0-42). Higher score indicate more insomnia
Bergen Insomnia Scale | 12 weeks after baseline.
  Self rated level of sleep problems. Range (0-42). Higher score indicate more insomnia
Bergen Insomnia Scale | 6 months after baseline.
  Self rated level of sleep problems. Range (0-42). Higher score indicate more insomnia
Beck depression Inventory II (Suicid item) | 8 weeks after baseline.
  Self reported level of suicidality. Range (0-3). Higher score indicate more suicidality.
Beck depression Inventory II (Suicid item) | 12 weeks after baseline.
  Self reported level of suicidality. Range (0-3). Higher score indicate more suicidality.
Beck depression Inventory II (Suicid item) | 6 months after baseline.
  Self reported level of suicidality. Range (0-3). Higher score indicate more suicidality.
Dot probe | 8 weeks after baseline.
  Degree of attentional bias- Measure mean reaction time.
Dot probe | 12 weeks after baseline
  Degree of attentional bias- Measure mean reaction time.
Dot probe | 6 months after baseline.
  Degree of attentional bias- Measure mean reaction time.
Facial Expression Rating Task | 8 weeks after baseline
  Measure of detection threshold for correctly identifying the emotional facial expression. Measures of number of correct answer (Range 0-100%)
Facial Expression Rating Task | 12 weeks after baseline
  Measure of detection threshold for correctly identifying the emotional facial expression. Measures of number of correct answer (Range 0-100%)
Facial Expression Rating Task | 6 months after baseline
  Measure of detection threshold for correctly identifying the emotional facial expression. Measures of number of correct answer (Range 0-100%)

CONTACTS AND LOCATIONS:
Overall Officials: Jan I Røssberg, PhD, Principal Investigator — Universitetet i Oslo/Oslo universitetssykehus
Locations (1):
- Jan Ivar Røssberg, Oslo, Nydalen, Norway

IPD SHARING:
Plan to Share IPD: Undecided
Anonymized data may be shared on request